CLINICAL TRIAL: NCT06163092
Title: The Prevalence of Chronic Endometritis and Therapeutic Benefits of Antibiotics in Women With Unexplained Recurrent Miscarriage
Brief Title: Chronic Endometritis and Benefits of Antibiotics in Women With Recurrent Miscarriage
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2023.526
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Miscarriage
Keywords: chronic endometritis; antibiotics; unexplained recurrent miscarriage women
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational study: Women with recurrent miscarriage would be invited to do endometrial sampling (ES) procedure. The ES will be conducted precisely 7 days after LH surge. It will be obtained using a Pipelle sampler as an outpatient procedure.

INTERVENTIONS:
Other:  — If the CE is high, antibiotics will be given to the patients as usual practice in hospitals.

SUMMARY:
The aim of the study is to estimate the incidence of CE, evaluate the endometrial microorganism of CE, and investigate the therapeutic benefits of antibiotics for women with unexplained recurrent miscarriage and CE.

DETAILED DESCRIPTION:
Eligible women, based on the inclusion and exclusion criteria, will be recruited from the miscarriage clinic in the Prince of Wales Hospital. Endometrial sampling (ES) will alternatively be conducted during mid-luteal phase. In natural cycles, all the subjects will have a daily urine test from day 9 of the menstrual cycle to identify the Luteinizing Hormone (LH) surge. The ES will be obtained precisely 7 days after LH surge. Endometrial samples will be obtained using a Pipelle sampler as an outpatient procedure. The endometrium will be divided into three aliquots. One will be fixed in 4% formalin for 24 hours, routinely processed and embedded in paraffin wax. One will be investigated by microbial culture for infectious agents and one will be sequenced to reveal the endometrial microbiota.

CE will be diagnosed either by the presence of plasma cells and changes in endometrial stromal cells identified using HE and IHC, or by the finding of infectious agents using microbial culture. The selection of antibiotics will be based on the type of infectious agents or empirical, doxycycline 100mg BD po. for 14 days, for women with negative microbial culture. Endometrial biopsy will be repeated at the same time point after antibiotic treatment for women with CE. For persistent subjects with negative culturing, ciprofloxacin 500mg, BD po., and metronidazole 400mg TDS po. for 14 days will be used. The treatment will be repeated for three courses at maximum for women with persistent CE according to their willingness.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of 2 or more consecutive miscarriages before 24 weeks of gestation
* Women aged 20-45 years old

Exclusion Criteria:

* Uncorrected uterine anomalies, such as the septate or bicornuate uterus, fibroids (submucous/intramural)
* Untreated hydrosalpinx
* Antiphospholipid syndrome
* Known clinical autoimmune disease
* Undergoing immunotherapy
* Abnormal thyroid function
* Abnormal karyotyping of couples
* Known immunodeficiency pathologies such as diabetes or HIV
* Currently taking other antibiotics or other trial medications or TCM;
* Currently or previously involved in other clinical trials with medication intake;
* Those with active pelvic inflammatory disease or suspicion of infection etc.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Please kindly see the inclusion criteria. The endometrics sampling is only done for female patients.
Study Population: Subjects will be identified and recruited from the miscarriage clinic by clinicians and research assistants and research nurse.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of chronic endometritis in local women with unexplained recurrent miscarriage | 31 January 2027
  the incidence of chronic endometritis in local women with unexplained recurrent miscarriage

SECONDARY OUTCOMES:
Investigate the spectrum of endometrial microorganisms associated with chronic endometritis in this population | 31 January 2027
  Investigate the spectrum of endometrial microorganisms associated with chronic endometritis in this population
Assess the clinical pregnancy outcomes between cured CE group and non-CE group | 31 January 2027
  Assess the clinical pregnancy outcomes in both cured CE group and non-CE group

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Pui Wah Chung, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No